CLINICAL TRIAL: NCT01603134
Title: A Randomized, Open Label, Two-Period, Two-Treatment, Two-Sequence, Single Dose, Crossover Comparative Bioequivalence Study of Allopurinol 300 mg Tablets USP With Zyloprim® 300 mg in Normal, Healthy, Adult, Human Male Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Allopurinol 300 mg Tablets USP Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IPCA Laboratories Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ipca/US/07/030
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Fasting State
MeSH Terms: interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol 300 mg Tablets USP (Experimental): Allopurinol 300 mg Tablets USP of M/s Ipca Laboratories Limited, India
  Interventions: Drug: Allopurinol
- Zyloprim® (Active Comparator): Zyloprim® (Allopurinol) 300 mg Tablets manufactured by Catalytica Pharma Inc., USA for Prometheus Laboratories Inc., USA,
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — 300 mg tablet once a day
  Other Names: Test Product
  Arms: Allopurinol 300 mg Tablets USP
Drug: Allopurinol — 300 mg tablet once a day
  Other Names: Zyloprim®
  Arms: Zyloprim®

SUMMARY:
This is a randomized, open Label, balanced, two-treatment, two-period, two-sequence, single dose, cross over comparative pivotal study. The purpose of this study is to assess the bioequivalence between Test Product and the corresponding Reference Product under fasting condition in normal, healthy, adult, human male subjects.

DETAILED DESCRIPTION:
Objective of this pivotal study was to assess the bioequivalence between Test Product: Allopurinol 300 mg Tablets USP of M/s Ipca Laboratories Limited, India and the corresponding Reference Product: Zyloprim® (Allopurinol) 300 mg Tablets manufactured by Catalytica Pharma Inc., USA for Prometheus Laboratories Inc., USA, under fasting condition in normal, healthy, adult, human male subjects in a randomized crossover study.

The study was conducted with 32 healthy adult male subjects. In each study period, a single 300 mg dose of either test or reference was administered to the subjects as per the randomization schedule in each study period with about 240 mL of water at ambient temperature in sitting position.

The duration of the clinical phase was 51 days including washout period of at 18 days between administrations of study drug in each study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects in the range of 18 - 45 years of age (Inclusive).
2. The healthy human male subjects, whose body weight within ± 15% of ideal weight as related to height and body frame according to Life Insurance Corporation (LIC) Chart.
3. Subjects with normal findings as determined by baseline history, physical examination and vital signs (blood pressure, pulse rate, respiration rate and oral temperature).
4. Subjects with normal findings, as determined by hematological tests, serum biochemistry, urine analysis, ECG and X-ray (if required).
5. Willingness to follow the protocol requirements as evidenced by written informed consent.
6. Agreeing to, not using any medication(either prescribed, OTC or alternate medicines), including vitamins and minerals for 14 days prior to study and during the course of the study.
7. No history or presence of significant alcoholism in the past one year.
8. Non-smokers, ex-smokers and light smokers will be included. "Light smokers are defined as someone smoking 10 cigarettes or less per day, ex-smokers as someone who completely stopped smoking for at least 3 months.

Exclusion Criteria:

1. Requiring medication for any ailment including enzyme-modifying drugs in the previous 28 days, before day one (1) of dosing.
2. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
3. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, hematological, gastrointestinal, endocrine, immunological or psychiatric diseases.
4. Subjects with history of recent myocardial infraction, cardiac arrhythmias, cardiac failure and convulsions.
5. Participation in a clinical drug study or bioequivalence study 90 days prior to present study.
6. History of malignancy or other serious diseases.
7. Refusal to abstain from food for at least ten (10.00) hours prior to administration of study drug and for at least four (04.00) hours post-dose.
8. Refusal to abstain from water for at least one (01.00) hour prior to study drug administration of each study period and for at least two (02.00) hours post-dose except about 240 mL administered during administration dose.
9. Any contraindication with blood sampling.
10. Refusal to abstain from smoking or consumption of tobacco products 48.00 hours before dosing until the last sample collection of each period.
11. Found positive in breath alcohol test done at the time of check-in for each study period.
12. History of drug abuse in past one year.
13. Use of xanthine-containing beverages or food, and fruit juice or grapefruit juice products for 48.00 hours prior to each drug dose.
14. Blood donation 90 days prior to the commencement of the study.
15. Subjects with positive HBsAg or Hepatitis-C, HIV tests and anti Treponema Palladium/Syphilis test.
16. History of hypersensitivity to Allopurinol or any ingredients of formulation.
17. History of problem in swallowing Tablet(s).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters. | 6 months
  Area Under Curve (AUC) and Cmax Sampling Hours: Pre-dose and at 00.25, 00.50, 00.75, 01.00, 01.25, 01.50, 01.75, 02.00, 02.25, 02.50, 02.75, 03.00, 03.50, 04.00, 04.50, 05.00, 05.50, 06.00, 06.50, 07.00, 08.00, 10.00, 12.00, 16.00, 24.00, 48.00, 72.00 and 96.00 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nirav Gandhi, M.D., Principal Investigator — Accutest Research Lab (I) Pvt. Ltd.
Locations (1):
- Accutest Research Lab (I) Pvt. Ltd., Ahmedabad, Gujarat, India